CLINICAL TRIAL: NCT04371952
Title: Doxycycline Versus Placebo in COVID-19 + Patients Without Hospitalization Criteria: Prospective, Multicenter, Randomized, Double-blind Study
Brief Title: DYNAMIC Study (DoxycYcliNe AMbulatoIre COVID-19)
Acronym: DYNAMIC
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: withdrawal due to the evolution of the epidemic, the arrival of vaccination and because the associated centres could no longer commit to the number of inclusions requested
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC20_0191
Record Dates: First submitted 2020-04-27; First posted 2020-05-01 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19 | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxycycline 100mg (Experimental): Doxycycline capsule containing 2 tablets doxycycline 100mg over-encapsulated. Doxycycline is given at 200 mg once a day and administered per os during 2 weeks
  Interventions: Drug: Doxycycline
- Doxycycline placebo (Placebo Comparator): Doxycycline Placebo capsule 200 mg, containing 1 capsule of a marketed placebo = RODAEL placebo ( lactose, 380 mg / capsule). Doxycycline placebo is given once a day and administered per os during 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline — comparison of doxycycline 200 mg/day to placebo
  Arms: Doxycycline 100mg
Drug: Placebo — Placebo : lactose, 380 mg/gélule
  Arms: Doxycycline placebo

SUMMARY:
The aim of the study is to compare a treatment with doxycycline vs a placebo as soon as the patient is confirmed COVID-19 + and before the onset of oxygen dependence with the aim of reducing or even abolishing the cytokine explosion and thus the evolution towards a serious form of the disease which can lead to death.

Three criteria support the rational use of tetrcycline in COVI-19 (1) The coronaviruses is known to bind to metalloproteases (MMPs) of the host, in particular to ensure viral survival. Tetracyclines are known to chelate zinc from MMPs. Their chelating activity may help inhibit COVID19 infection by limiting its ability to replicate in the host. (2) Tetracyclines may also be able to inhibit the replication of positive-polarity single-stranded RNA viruses, such as COVID19 (demonstrated on the dengue virus). (3) In addition, tetracyclines are modulators of innate immunity (anti-inflammatory activity), a property used in the treatment of inflammatory skin diseases for many years. These modulating effects are noted on several targets of innate immunity: They can decrease the expression of NFKB, the release of inflammatory cytokines such as TNF-α, IL-1β and IL-6, inhibit granulomas inflammatory and free radical release.

Tetracyclines could therefore participate in limiting the cytokine release induced by COVID19. Their lipophilic nature and their strong pulmonary penetration could allow them to inhibit viral replication.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman > 45 years old.
* Patient with a positive SARS-CoV-2 PCR
* Patient with ENT and / or respiratory symptoms, without hospitalization criteria (no dyspnea, respiratory rate <22 / min, SaO2 ≥ 94% in ambient air), or digestive signs.
* Patient with at least one of the following risk factors for unfavorable outcome:

  * 70 years, BMI> 30, cardiovascular history (stroke, coronary artery disease, complicated hypertension, cardiac surgery, NYHA III or IV heart failure), respiratory pathology likely to decompensate during viral infection respiratory failure, unbalanced and / or complicated diabètes, respiratory pathology likely to decompensate in the event of of viral infection, patients with renal insufficiency chronic dialysis, .cancer patients under treatment.

Exclusion Criteria:

* Lactose-intolerant patients
* Patient needing immediate hospitalization for any medical reason
* Patient having more than 5 days of clinical symptoms at the inclusion visit
* Patients with a history of allergy to tetracyclines
* Pregnant or lactating women
* Patients participating in another clinical trial
* Patients with photosensitive skin pathology
* Patients treated with anticoagulant
* Patients treated with oral retinoids: isotretinoin, alitretinoin, acitretin
* Patients treated with vitamin A Patients treated with systemic antibiotics for the duration of treatment
* Patients treated with barbiturates, carbamazepine or phenytoin
* Patients with treatment that may have an effect on COVID-19 infection: chloroquine, hydroxychloroquine, remdesivir, ganciclovir, acyclovir, ribavirin, lopinavir-ritonavir
* Patients under guardianship or trusteeship or in safeguard of justice

Min Age: 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients with Clinical Respiratory Aggravation | after at least 48 hours of treatment
  Percentage of patients with clinical worsening (SaO2 ≤ 93%) after at least 48 hours of treatment
Percentage of patients hospitalized | after at least 48 hours of experimental treatment
  Percentage of patients hospitalized after at least 48 hours of experimental treatment
Percentage of patients requiring ventilatory assistance | Day 0 to Day 28
  Percentage of patients requiring ventilatory assistance

SECONDARY OUTCOMES:
Positive SARS-CoV-2 PCR Test | Day -1 or day 0 AND Day 7
  Number of positive SARS-CoV-2 PCR tests on D-1 / D0 and D7 (+/- 2 days)
Duration of symptoms | Day 0 to Day 28
  Duration of symptoms (fever, painful symptoms: headache, sore throat, dyspnea)
Duration of hospitalization | From day 0 until to the end of hospitalization or date of death for any cause, whichever came first, assessed up to 3 months after Day0
  Total duration of hospitalization
Hospitalization intensive care or reanimation | From day 0 until to the end of hospitalization or date of death for any cause, whichever came first, assessed up to 3 months after Day0
  Duration of hospitalization in intensive care or reanimation
Duration of mechanical ventilatory assistance | to the end of mechanical ventilatory assistance if any, assessed up to 3 months after Day0
  Duration of mechanical ventilatory assistance
Percentage of deaths related to SARS-CoV-2 | Day 28, or end of hospitalization if any (assessed up to 3 months after Day0)
  Percentage of deaths related to SARS-CoV-2 infection
AE / SAE in both arms | Day 28, or end of hospitalization if any (assessed up to 3 months after Day0)
  Number of AE / SAE in both arms

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU Avicenne - APHP, Bobigny
  - CHU Bordeaux, Bordeaux
  - CHU Caen, Caen
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CHU Nantes, Nantes

IPD SHARING:
Plan to Share IPD: No